CLINICAL TRIAL: NCT01131546
Title: A Randomized, Controlled, Multicenter Trial of Levamlodipine Besylate Versus Amlodipine Maleate in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of Levamlodipine Besylate Compared to Amlodipine Maleate in Patients With Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Jinsheng Ren, Jiangsu Simcere Pharmaceutical R&D Co. Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM-77
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Levamlodipine Besylate; Amlodipine Maleate
MeSH Terms: conditions — Essential Hypertension | interventions — levamlodipine besylate; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levamlodipine besylate (2.5mg) (Experimental)
  Interventions: Drug: Levamlodipine besylate
- Levamlodipine besylate (5mg) (Experimental)
  Interventions: Drug: Levamlodipine besylate
- Amlodipine maleate (5mg) (Active Comparator)
  Interventions: Drug: Amlodipine maleate

INTERVENTIONS:
Drug: Levamlodipine besylate — Once daily, 7AM - 10AM
  Arms: Levamlodipine besylate (2.5mg); Levamlodipine besylate (5mg)
Drug: Amlodipine maleate — Once daily, 7AM - 10AM
  Arms: Amlodipine maleate (5mg)

SUMMARY:
This study is designed to compare the safety and efficacy of levamlodipine besylate (2.5mg or 5mg) versus amlodipine maleate (5mg) in patients with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, 18-75 Years
* Patients with mild to moderate essential hypertension (defined as mean BP of 2 visits ≥140mm/90mmHg, and < 180mm/110mmHg)
* Written informed consent

Exclusion Criteria:

* Patients with secondary hypertension
* Patients with severe hypertension
* Have to take other drugs that can influence blood pressure during the study
* Allergic to DHP calcium antagonists
* Evidence of congestive heart failure, unstable angina or severe arrhythmia
* Renal or hepatic dysfunction
* Women who are taking contraceptive pills or are likely to be pregnant
* Participate in other clinical trials within 3 months prior to this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who reach overall blood pressure control (defined as BP <140/90 mmHg for non-diabetic patients and < 130/80 mmHg for diabetic patients) | Week 8

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure (SBP) | Week 8
Change from baseline in diastolic blood pressure (DBP) | Week 8
Incidence of adverse effects | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dayi Hu, MD, Principal Investigator — Peking University People's Hospital; Jinming Yu, Ph.D., Principal Investigator — School of Public Health，Fudan University
Locations (1):
- Peking University People's Hospital, Beijing, China